Clinical Efficacy Analysis of Resveratrol in the Treatment of

**Primary Ovarian Insufficiency** 

Date: May 16, 2022

**Research Proposal Summary** 

Statistical analysis

The case observation form completed by the test center was reviewed and

returned by the project team of Reproductive Medicine Center, Affiliated

Hospital of Nantong University, and the data was processed by a

statistical analyst. The data in the case report form is entered in two

copies, and the database is locked after verification and confirmation.

SPSS26.0 software was used for statistical analysis. The full analysis set

(FAS) and the per-protocol set (PPS) were used for effectiveness analysis,

and the safety data set (SS) was used for safety analysis. Measurement

data were expressed as mean±standard deviation ( $\bar{x}\pm s$ ), multiple time

points were compared by repeated measures analysis of variance, and

pairwise comparisons were by Bonferroni test; enumeration data were

expressed by the number of cases or percentages, and  $\chi^2$  was used. Test

for statistical comparison. P<0.05 indicated that the difference was

statistically significant.